CLINICAL TRIAL: NCT00919672
Title: Treatment of Irritable Bowel Syndrome (IBS) With Sacral Nerve Stimulation. A Blinded, Randomized Crossover Study
Brief Title: Treatment of Irritable Bowel Syndrome (IBS) With Sacral Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070218,JLF
Record Dates: First submitted 2009-05-25; First posted 2009-06-12 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Sacral nerve stimulation; Motility; Pain perception; GSRS-IBS; IBS-IS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sacral nerve stimulation ON-OFF (Active Comparator): As previously described the patients will be randomized in a blinded design to receive either ON-OFF or OFF-ON stimulation in a 2 month period.
  Interventions: Device: Sacral nerve stimulation
- Sacral nerve stimulation OFF-ON (Active Comparator): As previously described the patients will be randomized in a blinded design to receive either ON-OFF or OFF-ON stimulation in a 2 month period.
  Interventions: Device: Sacral nerve stimulation

INTERVENTIONS:
Device: Sacral nerve stimulation — The stimulation is set individually to provide the best possible stimulation for each individual person. This setting is found before the study starts and will not be altered during the study.
  Other Names: Irritable Bowel Syndrome

SUMMARY:
Sacral nerve stimulation (SNS) has become a well-established treatment for patients with fecal incontinence since 1995. The mechanism of action of SNS is still not fully understood but recent studies have shown that the motility of the whole colon is modulated during the stimulation. This modulation of the colonic motility could be a potential mechanism of an action to relieve the symptoms in patients with IBS.

Twenty eight patients with IBS will be enrolled in the study. They have to meet the ROME III criteria, and also satisfy the criteria for implantation of a neurostimulator.

After a post implantation period where the programming of the neurostimulator is optimised, the patient is randomized in a double blinded design to receive either ON-OFF or OFF-ON stimulation in a 2-month period.

At the end of each period (ON/OFF) the patient will be examined with Magnet Tracking System (MTS) for motility and with impedance planimetry including thermal stimulation (circulating water)for multimodal sensory testing of the rectum.

This is based on the study hypothesis that the motility of the small intestine and the colon is changed in IBS patients according to their subtype (Diarrhoea-IBS, Constipation-IBS and Disordered bowel habit-IBS) compared to healthy persons. And that SNS will affect the motility of the small intestine and the colon in IBS patients as well as SNS will affect the perception of pain/discomfort in the rectum in IBS patients.

The effect of ON-OFF-sacral nerve stimulation on the IBS patients and thereby their IBS symptoms will also be evaluated by an IBS score (GSRS-IBS)and on quality of life by an IBS Impact Scale (IBS-IS) as well as the significance of placebo effect in the treatment of patients with IBS with SNS will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Patients who are psychologically stable and suitable for intervention and able to provide informed consent.
* Patients who are diagnosed with IBS according to the Rome III criteria
* Minimum 30% reduction of the IBS symptoms during the PNE-test (a criteria for implantation of the neurostimulator)

Exclusion Criteria:

* Overt bowel diseases including inflammatory bowel disease
* Pregnant or breast feeding
* Patients who are considered unable to follow the planned programme of the study, including mentally illness or physiological instability
* Patients who are on medication with known influence on gastrointestinal motility including those for thyroid disease, diabetes mellitus, celiac disease and neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Comparing the investigations with MTS and impedance planimetry as well as the GSRS-IBS and IBS-IS scores in the the two periods (ON/OFF periods) in the single IBS patient. Nonparametrics tests. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lilli Lundbye, PhD, Study Director — Analfysiologisk Klinik, University Hospital of Aarhus
Locations (1):
- Analfysiologisk Klinik, University Hospital of Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Fassov J, Lundby L, Worsoe J, Buntzen S, Laurberg S, Krogh K. A randomised, controlled study of small intestinal motility in patients treated with sacral nerve stimulation for irritable bowel syndrome. BMC Gastroenterol. 2014 Jun 25;14:111. doi: 10.1186/1471-230X-14-111. PMID 24965754